CLINICAL TRIAL: NCT02328027
Title: A Phase I-IIa Study of Safety, Tolerance, Pharmacokinetics, Dosimetry and Benefice of Early Nuclear Medicine Imaging of 99mTc-rhAnnexin V-128 in Patients With Rheumatoid Arthritis or Ankylosing Spondylitis
Brief Title: 99mTc-rhAnnexin V-128 a Phase I/IIa Study in Patients With Rheumatoid Arthritis (RA) or Ankylosing Spondylitis (AS)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Low recruitment
Sponsor: Advanced Accelerator Applications (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1002; CAAA113A22101 (Other: Novartis)
Record Dates: First submitted 2014-12-18; First posted 2014-12-31 (Estimated); Results first posted 2020-06-09 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-09

CONDITIONS: Rheumatoid Arthritis; Ankylosing Spondylitis
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylitis, Ankylosing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 99mTc-rhAnnexin V-128, i.v. (Experimental): Patients will receive 2 administrations of the 99mTc-rhAnnexin V-128 medical imaging agent: one at Day 1 and the other at Day 42.
  Interventions: Drug: 99mTc-rhAnnexin V-128

INTERVENTIONS:
Drug: 99mTc-rhAnnexin V-128 — 1 single intravenous bolus administration of 250 MBq, at Day 1 and at Day 42.

SUMMARY:
This was a monocentric, open label, Phase I-IIa study. Eligible patients who signed the ICF received two single intravenous (IV) bolus of the imaging agent 99mTc-rhAnnexin V-128. The first dose was administered on Day 1, and the second dose on Day 42 (±2 weeks).

All patients were to start a new disease modifying treatment for RA or AS on Day 2. This disease modifying treatment was at the discretion of the investigator and was not chosen by the sponsor.

Safety was monitored at every visit. Whole body scintigraphic imaging was performed at Day 1 and Day 42 after 99mTc-rhAnnexin V-128 dosing. Clinical disease assessments were performed at screening, Day 42 and Day 90 to assess response to RA or AS treatment. Blood was drawn to test for 99mTc-rhAnnexin V-128 immunogenicity at screening and on Days 30, 56 and 90. Patients participating in the pharmacokinetic (PK)/dosimetric sub-study had additional assessments in the 24 hours following the Day 1 dose of 99mTc-rhAnnexin V-128.

DETAILED DESCRIPTION:
The study was terminated early after the inclusion of 16 of the 20 planned patients. The sponsor decided to terminate the study earlier than planned due to slow accrual. Novartis acquired Advanced Accelerator Applications SA.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with RA based on ACR/EULAR 2010 criteria (score >=6), or Patients diagnosed with AS based on the ASAS criteria. Patients with RA must have serology assessment performed and documented at the time of enrollment.
* Patient with RA active disease (DAS > 2,6) and the introduction of a Bi-DMARD should be indicated. RA patients must have been treated with DMARD (methotrexate, leflunomide and sulfasalazine) or combination of these treatments for at least 3 months. Treatment will be pursued while on study.

or RA patients must have been previously treated with Bi-DMARD before initiation of the new Bi-DMARD treatment. The non-response of the previous Bi-DMARD treatment must be documented.

or Patients with AS with insufficiently controlled disease while under NSAID and indication for Bi-DMARD. These patients must be under NSAID for at least 3 months and under the same NSAID for at least 1 month prior to enrollment.

* ≥ 18 years old
* Karnofsky ≥ 80%
* Negative Pregnancy test for women with childbearing potential
* For women with childbearing potential, use of two reliable means of contraception (e.g., hormonal contraceptive, patch, vaginal ring, intrauterine device, associated with other barrier method of contraception such as the use of condoms) , throughout their participation in the study
* Absence of ECG anomaly
* written ICF signed

Exclusion Criteria:

* Pregnancy or lactation
* Liver impairment (ALT, AST or Bilirubin > 2 ULN) at screening visit or baseline
* Kidney impairment (serum creatinine > 1.5 mg/dL)
* History of congestive heart failure (NYHA III & IV)
* History of malignant disease within 5 years
* History of any disease or relevant physical or psychiatric condition or abnormal physical finding which may interfere with the study objectives at the investigator judgment
* Known hypersensitivity to the investigational drug or any of its components
* Participation to another clinical trial within 4 weeks before study inclusion except for patients who have participated or who are currently participating in an interventional study without any study drug administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-12-11 (Actual); Primary Completion 2017-10-17 (Actual); Study Completion 2017-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Prior, MD, PhD, Principal Investigator — CHUV Lausanne; Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: It was planned that 20 evaluable patients with either RA or AS (enrolled in a 1:1 ratio) would be included and would complete the assessments on Day 56, however recruitment was terminated after inclusion of 16 patients.
Pre-assignment Details: Of the 16 enrolled participants, 10 participants would take part in a PK/dosimetric sub-study, after providing written approval (only 5 participants were enrolled to the sub-study). Of the first 6 enrolled participants overall, at least 3 had to take part in the sub-study to optimise the PK time points for subsequent participants .
Groups:
- 99mTc-rhAnnexin V-128: Ankylosing Spondylitis: Participants with Ankylosing Spondylitis (AS) received a single bolus injection of 99mTc-rhAnnexin V-128 at a dose of 250 Megabecquerel (MBq) through an intravenous (IV) catheter in an antecubital vein, followed by a saline flush on Day 1 and on Day 42.
- 99mTc-rhAnnexin V-128: Rheumatoid Arthritis: Participants with Rheumatoid Arthritis (RA) received a single bolus injection of 99mTc-rhAnnexin V-128 at a dose of 250 MBq through an IV catheter in an antecubital vein, followed by a saline flush on Day 1 and on Day 42.
Period: Overall Study
Arm/Group | 99mTc-rhAnnexin V-128: Ankylosing Spondylitis | 99mTc-rhAnnexin V-128: Rheumatoid Arthritis
Started | 5 | 11
Completed | 5 | 10
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set included participants who have received at least one dose of study drug.
Groups:
- 99mTc-rhAnnexin V-128: Ankylosing Spondylitis: Participants with AS received a single bolus injection of 99mTc-rhAnnexin V-128 at a dose of 250 MBq through an IV catheter in an antecubital vein, followed by a saline flush on Day 1 and on Day 42.
- 99mTc-rhAnnexin V-128: Rheumatoid Arthritis: Participants with RA received received a single bolus injection of 99mTc-rhAnnexin V-128 at a dose of 250 MBq through an IV catheter in an antecubital vein, followed by a saline flush on Day 1 and on Day 42.
- Total: Total of all reporting groups
Arm/Group | 99mTc-rhAnnexin V-128: Ankylosing Spondylitis | 99mTc-rhAnnexin V-128: Rheumatoid Arthritis | Total
Number analyzed (Participants) | 5 | 11 | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.2 (10.73) | 51.6 (18.74) | 49.0 (16.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 9 | 9
  Male | 5 | 2 | 7
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 4 | 11 | 15
  Hispanic | 1 | 0 | 1
Region of Enrollment [Number; unit: Participants]
  Switzerland | 5 | 11 | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events (SAE) and Death
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient and which does not necessarily have a causal relationship with the study medication. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease, temporally associated with the use of a study medication, whether or not causally related to the study medication. TEAEs are defined as all AEs reported after the first dose. An SAE is any untoward medical occurrence that at any dose: results in death, is life-threatening, life-threatening, results in persistent or significant disability/incapacity, results in congenital anomaly or birth defect, requires in-patient hospitalization or leads to prolongation of hospitalization.
Time Frame: From screening up to Day 90
Population: Safety analysis set included all participants who have received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- 99mTc-rhAnnexin V-128: Ankylosing Spondylitis: Participants with AS received received a single bolus injection of 99mTc-rhAnnexin V-128 at a dose of 250 MBq through an IV catheter in an antecubital vein, followed by a saline flush on Day 1 and on Day 42.
- 99mTc-rhAnnexin V-128: Rheumatoid Arthritis: Participants with RA received a single bolus injection of 99mTc-rhAnnexin V-128 at a dose of 250 MBq through an IV catheter in an antecubital vein, followed by a saline flush on Day 1 and on Day 42.
Arm/Group | 99mTc-rhAnnexin V-128: Ankylosing Spondylitis | 99mTc-rhAnnexin V-128: Rheumatoid Arthritis
Number analyzed (Participants) | 5 | 11
Participants
  TEAEs | 3 | 11
  SAEs | 0 | 1
  Death | 0 | 0

2. Secondary Outcome: Area Under the Curve Extrapolated to Infinity (AUC) of 99mTc-rhAnnexin V-128
Description: AUC is defined as area under the curve extrapolated to infinity of 99mTc-rhAnnexin V-128.
Time Frame: Day 1 (0 (Predose), 0.05, 0.10, 0.15, 0.30, 1.00, 1.50, 2.00, 4.00 and 24.00 hours)
Population: PK population included all participants who participated in the PK/dosimetry sub-study which included participants regardless of their diagnosis (RA or AS). Here 'n' (number analyzed) signifies participants who were evaluable for specified categories.
Measure: Mean (Standard Deviation); unit: nanogram*hour per milliliter (ng.h/mL)
Groups:
- 99mTc-rhAnnexin V-128: AS and RA: Participants with AS and RA received a single bolus injection of 99mTc-rhAnnexin V-128 at a dose of 250 MBq through an IV catheter in an antecubital vein, followed by a saline flush on Day 1 and on Day 42.
Arm/Group | 99mTc-rhAnnexin V-128: AS and RA
Number analyzed (Participants) | 5
nanogram*hour per milliliter (ng.h/mL)
  Blood: number analyzed (Participants) | 4
  Blood | 41.2 (13.7)
  Serum | 53.6 (22.6)

3. Secondary Outcome: Distribution Volume (Vz) of 99mTc-rhAnnexin V-128
Description: Vz is defined as the distribution volume of 99mTc-rhAnnexin V-128.
Time Frame: Day 1 (0 (Predose), 0.05, 0.10, 0.15, 0.30, 1.00, 1.50, 2.00, 4.00 and 24.00 hours)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Liters (L)
Arm/Group | 99mTc-rhAnnexin V-128: AS and RA
Number analyzed (Participants) | 5
Liters (L)
  Blood: number analyzed (Participants) | 4
  Blood | 30.3 (9.0)
  Serum | 26.1 (11.5)

4. Secondary Outcome: Systemic Clearance (Cl) of 99mTc-rhAnnexin V-128
Description: Cl is defined as the systemic clearance of 99mTc-rhAnnexin V-128.
Time Frame: Day 1 (0 (Predose), 0.05, 0.10, 0.15, 0.30, 1.00, 1.50, 2.00, 4.00 and 24.00 hours)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Liter per hour (L/h)
Arm/Group | 99mTc-rhAnnexin V-128: AS and RA
Number analyzed (Participants) | 5
Liter per hour (L/h)
  Blood: number analyzed (Participants) | 4
  Blood | 5.82 (1.59)
  Serum | 4.68 (1.67)

5. Secondary Outcome: Elimination Half-life (t1/2) of 99mTc-rhAnnexin V-128
Description: t1/2 is defined as the elimination half-life of 99mTc-rhAnnexin V-128.
Time Frame: Day 1 (0 (Predose), 0.05, 0.10, 0.15, 0.30, 1.00, 1.50, 2.00, 4.00 and 24.00 hours)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 99mTc-rhAnnexin V-128: AS and RA
Number analyzed (Participants) | 5
hours
  Blood: number analyzed (Participants) | 4
  Blood | 3.6 (0.2)
  Serum | 3.8 (0.3)

6. Secondary Outcome: Serum Concentration of rhAnnexin V-128 Based on Enzyme-linked Immunosorbent Assay (ELISA) Analysis
Description: Serum concentration of rhAnnexin V-128 based on ELISA analysis were to be evaluated and reported overtime.
Time Frame: Day 1 (0 (Predose), 0.05, 0.10, 0.15, 0.30, 1.00, 1.50, 2.00, 3.00, 4.00, 6.00 and 24.00 hours)
Population: Pharmacokinetic (PK) population included all participants who participated in the PK/dosimetry sub-study which included participants regardless of their diagnosis (RA or AS). Due to low concentration of the protein in serum PK parameters could not be derived.
Arm/Group | 99mTc-rhAnnexin V-128: AS and RA
Number analyzed (Participants) | 0

7. Secondary Outcome: 99mTc-rhAnnexin V-128 Blood Cpm Decay Corrected Data (Counts Per Minute in 1 mL Sample)
Description: Total radioactivity count per minute in whole blood samples were reported.
Time Frame: Day 1 (0 (Predose), 0.05, 0.10, 0.15, 0.30, 1.00, 1.50 to 2.00, 3.00 to 4.00 and 24.00 hours)
Population: PK population included all participants who participated in the PK/dosimetry sub-study which included participants regardless of their diagnosis (RA or AS). Here 'n' (number analyzed) signifies participants who were evaluable at specified timepoints.
Measure: Mean (Standard Deviation); unit: counts per minute (CPM) in 1 mL sample
Arm/Group | 99mTc-rhAnnexin V-128: AS and RA
Number analyzed (Participants) | 5
counts per minute (CPM) in 1 mL sample
  0 (Predose): number analyzed (Participants) | 4
  0 (Predose) | 0.0 (0.00)
  5 min: number analyzed (Participants) | 4
  5 min | 1667814 (209478)
  10 min: number analyzed (Participants) | 4
  10 min | 1188917 (162265)
  15 min: number analyzed (Participants) | 4
  15 min | 976977 (168240)
  30 min: number analyzed (Participants) | 4
  30 min | 560111 (183995)
  1h: number analyzed (Participants) | 4
  1h | 270715 (101320)
  1.5h to 2.0h: number analyzed (Participants) | 4
  1.5h to 2.0h | 140730 (30842)
  3.0h to 4.0h: number analyzed (Participants) | 3
  3.0h to 4.0h | 64421 (20850)
  24h: number analyzed (Participants) | 4
  24h | 1803 (641)

8. Secondary Outcome: 99mTc-rhAnnexin V-128 Serum Cpm Decay Corrected Data (Counts Per Minute in 1 mL Sample)
Description: Total radioactivity count per minute in serum samples were reported.
Time Frame: Day 1 (0 (Predose), 0.05, 0.10, 0.15, 0.30, 1.00, 1.50 to 2.00, 3.00 to 4.00, 6.00 and 24.00 hours)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: counts per minute (CPM) in 1 mL sample
Arm/Group | 99mTc-rhAnnexin V-128: AS and RA
Number analyzed (Participants) | 5
counts per minute (CPM) in 1 mL sample
  Predose | 0.0 (0.00)
  5 min | 2043946 (654557)
  10 min | 1432102 (453282)
  15 min | 1176933 (299437)
  30 min | 719880 (287310)
  1h | 349309 (103963)
  1.5h to 2.0h | 223067 (51303)
  3.0h to 4.0h: number analyzed (Participants) | 4
  3.0h to 4.0h | 106070 (31082)
  6h: number analyzed (Participants) | 1
  6h | 56768 (NA) — NA: Not estimable due to the number of participants with events.
  24h | 3126 (1010)

9. Secondary Outcome: 99mTc-rhAnnexin V-128 Urine Cpm Decay Corrected Data (Counts Per Minute in 1 mL Sample)
Description: Total radioactivity count per minute in urine samples were reported.
Time Frame: Day 1 (0 (Predose), 1.00, 4.00, 6.00 and 24.00 hours)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: counts per minute (CPM) in 1 mL sample
Arm/Group | 99mTc-rhAnnexin V-128: AS and RA
Number analyzed (Participants) | 5
counts per minute (CPM) in 1 mL sample
  0 (Predose) | 12 (26)
  1 hour: number analyzed (Participants) | 3
  1 hour | 6613620 (1786521)
  4 hours | 9135076 (3248412)
  16 hours | 1517263 (1180019)
  24 hours | 96155.2 (84394.79)

10. Secondary Outcome: Number of Annexin Related Species as Assessed Size-Exclusion HPLC- High-Performance Liquid Chromatography (SEC-HPLC) Analysis
Description: Urine samples (10 mL aliquots) were analysed as a function of time by SEC-HPLC technique at the local laboratory in order to gain information on the chemical status of 99mTc-rhAnnexin V-128 and on the presence of 99mTc-rhAnnexin V-128-related species.
Time Frame: Day 1 (0 (Predose), up to 1.00 hour, from 1.00 to 4.00 hours, from 4.00 to 6.00 hours, from 16.00 to 24.00 hours)
Population: PK population included all participants who participated in the PK/dosimetry sub-study which included participants regardless of their diagnosis (RA or AS).
Measure: Count of Participants; unit: Participants
Arm/Group | 99mTc-rhAnnexin V-128: AS and RA
Number analyzed (Participants) | 5
Participants
  0 (Predose)-HPLC Performed?=Yes: Species found = No | 5
  0 (Predose)-HPLC Performed?=Yes: Species found = Not Specified | 0
  Up to 1 hour-HPLC Performed?=Yes: Species found = No | 5
  Up to 1 hour-HPLC Performed?=Yes: Species found = Not Specified | 0
  From 1 to 4 hours-HPLC Performed?=Yes: Species found = No | 5
  From 1 to 4 hours-HPLC Performed?=Yes: Species found = Not Specified | 0
  From 4 to 6 hours-HPLC Performed?=Yes: Species found = No | 5
  From 4 to 6 hours-HPLC Performed?=Yes: Species found = Not Specified | 0
  From 16 to 24 hours-HPLC Performed?=Yes: number analyzed (Participants) | 4
  From 16 to 24 hours-HPLC Performed?=Yes: Species found = No | 4
  From 16 to 24 hours-HPLC Performed?=Yes: Species found = Not Specified | 0
  From 16 to 24 hours-HPLC Performed?=No: number analyzed (Participants) | 1
  From 16 to 24 hours-HPLC Performed?=No: Species found = No | 0
  From 16 to 24 hours-HPLC Performed?=No: Species found = Not Specified | 1

ADVERSE EVENTS:
Time Frame: From start of screening up to Day 90
Description: Safety set included all eligible participants who were administered at least one treatment.
Arm/Group | 99mTc-rhAnnexin V-128: Ankylosing Spondylitis | 99mTc-rhAnnexin V-128: Rheumatoid Arthritis
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/5 | 1/11
Other Adverse Events (participants affected / at risk) | 3/5 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 99mTc-rhAnnexin V-128: Ankylosing Spondylitis (N=5) | 99mTc-rhAnnexin V-128: Rheumatoid Arthritis (N=11)
Depression (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 99mTc-rhAnnexin V-128: Ankylosing Spondylitis (N=5) | 99mTc-rhAnnexin V-128: Rheumatoid Arthritis (N=11)
Angina pectoris (Cardiac disorders) | 0 | 1
Cyanosis (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1
Faeces discoloured (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1
Chills (General disorders) | 0 | 1
Fatigue (General disorders) | 2 | 4
Influenza like illness (General disorders) | 0 | 2
Malaise (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 2
Cytokine release syndrome (Immune system disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 1
Procedural dizziness (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Blood urine present (Investigations) | 0 | 1
Oxygen saturation decreased (Investigations) | 0 | 1
Weight decreased (Investigations) | 0 | 1
Weight increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 1
Dementia (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 3
Paresis (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Urinary tract pain (Renal and urinary disorders) | 0 | 1
Urine odour abnormal (Renal and urinary disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The sponsor decided to terminate the study earlier than planned due to slow accrual (16 of the planned 20 patients).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2014-12-16): https://cdn.clinicaltrials.gov/large-docs/27/NCT02328027/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-26): https://cdn.clinicaltrials.gov/large-docs/27/NCT02328027/SAP_001.pdf